CLINICAL TRIAL: NCT07339826
Title: Overview of Knowledge and Practices Among Healthcare Professionals Treating Eating Disorders in the Perinatal Context in Alsace, France
Brief Title: Overview of Knowledge and Practices Among Healthcare Professionals Treating Eating Disorders
Acronym: TCA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9769
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Eating Disorders
Keywords: Eating Disorders; Perinatal psychiatry
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perinatal psychiatry is a psychiatric specialty that has been developing for several years. This perinatal period is crucial for bio-psycho-affective development.

Eating disorders are among the most common disorders in psychiatry. Women who have experienced or currently experience eating disorders may exhibit a relapse, stabilization, or improvement in these behaviors, with direct consequences for their baby's development.

Although eating disorders have been extensively studied in adolescents and adults, the perinatal period remains less explored.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatrists, midwives, gynecologists, general practitioners, psychologists, maternal and child health professionals (PMI),
* Practicing in Alsace
* Agreeing to participate in the survey

Exclusion Criteria:

* Healthcare professionals who do not treat patients in a perinatal context.
* Professionals outside Alsace

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatrists, midwives, gynecologists, general practitioners, psychologists, maternal and child health professionals (PMI) practicing in Alsace
Sampling Method: Non-Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
Overview of healthcare professionals' practices concerning eating disorders in the perinatal period | Up to 12 months
  The study consists of an overview of healthcare professionals' practices concerning eating disorders in the perinatal period in the Alsace region of France

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Psychothérapique pour Enfants et Adolescents - CHU de Strasbourg - France, Strasbourg, France